CLINICAL TRIAL: NCT02971072
Title: Neurophysiology of Weakness and Exercise in Rotator Cuff Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05022014.005; 1R01AR063713-01A1 (NIH)
Record Dates: First submitted 2016-05-10; First posted 2016-11-22 (Estimated); Last update posted 2022-09-13 (Actual); Status verified 2020-03

CONDITIONS: Acute Pain; Atrophic; Goals; Impairment; Infiltration; Injury; Muscle Weakness; Pain; Pathology; Shoulder Pain; Syndrome; Tendinopathy
Keywords: address; atrophic; base; clinical; cost; data; disability; effectiveness; attention; biofeedback; electrical stimulation; electromyography; exercise; exertion; health care service utilization; improved; injection of therapeutic agent; innovation; intervention; knowledge; local anesthetics; measures; modeling; motor; motor control; muscle; neuroadaptation; neurophysiology; novel; outcome; outcome measure; pain inhibition; patients; pattern; programs; public health relevance; rehabilitation strategy; relating to nervous system; reporting; research; rotator cuff; shoulder; staging; strength training; success; systematic review; techniques; testing; time; training; treatment strategy; United States; work
MeSH Terms: conditions — Acute Pain; Atrophy; Wounds and Injuries; Muscle Weakness; Pain; Shoulder Pain; Syndrome; Tendinopathy; Motor Activity; Patient Acceptance of Health Care | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients (Experimental): Subjects with shoulder tendinopathy who will undergo both a subacromial injection and physical therapy
  Interventions: Procedure: Subacromial injection; Other: Physical Therapy

INTERVENTIONS:
Procedure: Subacromial injection — A subacromial injection consisting up 6 cc 0.5% Marcaine with Epinephrine and 1 cc DepoMedrol will be administered.
Other: Physical Therapy — A standardized six-week exercise protocol supervised by a physical therapist

SUMMARY:
The purpose of this study is to examine deficits in activation and motor patterns, as well as central drive in patients with rotator cuff tendinopathy. There are three specific aims: (1) determine the effect of acute pain relief on rotator cuff muscle activation in patients with rotator cuff tendinopathy, (2) determine the effect of exercise on rotator cuff muscle activation in patients with rotator cuff tendinopathy, and (3) compare rotator cuff muscle activation between patients with rotator cuff tendinopathy and healthy controls.

DETAILED DESCRIPTION:
The long-term goal of our research agenda is to identify the mechanisms associated with rotator cuff tendinopathy (impingement syndrome) and subsequently evaluate novel treatment strategies that address these mechanisms. The objectives of this application are to study the muscle patterns in patients with rotator cuff tendinopathy as well as the effects of both pain and exercise on these patterns. Our first hypothesis is that pain relief from a shoulder injection will result in increased rotator cuff activity. Our second hypothesis is that patients with tendinopathy will demonstrate improved rotator cuff muscle activity following a six-week exercise program and that this improvement will be higher in patients that respond favorably to treatment. Our final hypothesis is that patients with cuff tendinopathy will show decreased rotator cuff activity compared to healthy subjects. The investigators plan on addressing these hypotheses using several novel techniques for muscle activity assessment.

ELIGIBILITY:
Patient Inclusion Criteria:

* pain with passive provocative maneuvers (positive Hawkins or Neer test)
* pain with active elevation (positive painful arc)
* pain with isometric resisted movements (Jobe's "empty can" test or resisted shoulder external rotation with the arm at the side)
* demonstrate weakness (>10% force deficit in external rotation)

Patient Exclusion Criteria:

* shoulder surgery on the symptomatic side
* positive Spurling test
* traumatic shoulder dislocation or instability in the past 3 months
* reproduction of shoulder pain with active or passive cervical range of motion
* signs of rotator cuff tear (drop-arm test, lag signs, gross external rotation weakness, or positive image findings)
* current musculoskeletal, neurologic or cardiovascular compromise

Control Inclusion Criteria:

* no current or previous shoulder injury
* matched for age (within 5 years) and sex
* meet Patient Exclusion Criteria (minus musculoskeletal, neurologic, or cardiovascular compromise)

Control Exclusion Criteria:

* pain with active arm elevation
* positive Hawkins, Neer, or Jobe's test

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Rotator cuff activation after subacromial injection and exercise intervention, difference in rotator cuff voluntary activation between subjects and controls | 6 weeks
  Assessed using voluntary activation
Rotator cuff activation after subacromial injection and exercise intervention, difference in specific rotator cuff muscle activation between subjects and controls | 6 weeks
  Assessed using electromyography (EMG)

SECONDARY OUTCOMES:
Rotator cuff voluntary activation after subacromial injection | 2 hours
  Assessed using voluntary activation
Rotator cuff muscle activation after subacromial injection | 2 hours
  Assessed using EMG
Rotator cuff voluntary activation correlations with pain levels | 2 hours
  Assessed using voluntary activation relative to self-reported pain level
Rotator cuff activation correlations with pain levels | 2 hours
  Assessed using EMG relative to self-reported pain level
Rotator cuff voluntary activation after 6-week exercise intervention and subacromial injection | 6 weeks
  Assessed using voluntary activation
Rotator cuff muscle activation after 6-week exercise intervention and subacromial injection | 6 weeks
  Assessed using EMG
Rotator cuff voluntary activation correlation with improvements in pain relief | 6 weeks
  Assessed using voluntary activation relative to self-reported pain relief
Rotator cuff voluntary activation correlation with improvements in clinical outcome measures | 6 weeks
  Assessed using voluntary activation relative to changes in questionnaire scores
Rotator cuff muscle activation correlation with improvements in pain relief | 6 weeks
  Assessed using EMG relative to self-reported pain relief
Rotator cuff muscle activation correlation with improvements in clinical outcome measures | 6 weeks
  Assessed using EMG relative to changes in questionnaire scores
Prior to treatment, rotator cuff voluntary activation in patients relative to healthy controls | 6 weeks
  Assessed using voluntary activation
Prior to treatment, rotator cuff muscle activation in patients relative to healthy controls | 6 weeks
  Assessed using EMG
After both a subacromial injection and a six-week exercise program, differences in rotator cuff voluntary activation between patients and healthy controls | 6 weeks
  Assessed using voluntary activation
After both a subacromial injection and a six-week exercise program, differences in rotator cuff muscle activation between patients and healthy controls | 6 weeks
  Assessed using EMG

CONTACTS AND LOCATIONS:
Overall Officials: Andrew R Karduna, PhD, Principal Investigator — University of Oregon
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No